CLINICAL TRIAL: NCT01998802
Title: A Multi-Center, Double-Masked, Randomized, Controlled, Efficacy and Safety Study of EBI-005 5 mg/mL Topical Ophthalmic Solution Versus Vehicle Contraol In Subjects With Moderate to Severe Dry Eye Disease
Brief Title: Phase 3 Study of EBI-005 in Dry Eye Disease
Acronym: EBI-005
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBI-005-3
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator: EBI-005 (Active Comparator): Drug: EBI-005 The investigational drug EBI-005, is an intervention to one of two study arms: 5 mg/mL topical administered 3 times per day.
  Interventions: Drug: Active Comparator EBI-005
- Placebo Comparator (Placebo Comparator): One of two study arms: placebo topical administered 3 times per day.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Active Comparator EBI-005
  Arms: Active Comparator: EBI-005
Drug: Placebo Comparator
  Arms: Placebo Comparator

SUMMARY:
This is a phase III double-masked, randomized, controlled study evaluating the efficacy of EBI-005 as compared to vehicle given as a topical ophthalmic solution in each eye to subjects with moderate to severe DED three times daily for 12 weeks. Approximately 730 subjects at up to approximately 50 centers in the United States will be screened, enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and any authorizations required by local law (e.g., Protected Health Information waiver) prior to performing any study procedures;
* Are ≥ 18 years of age;
* Are willing and able to follow instructions and can be present for the required study visits for the duration of the study;
* Have a history of dry eye disease (DED) in both eyes supported by a previous clinical diagnosis
* Have normal lid anatomy.
* If female and of child bearing potential, she must not be not pregnant or lactating and not sexually active (abstinent) within 14 days prior to Visit 1

Exclusion Criteria:

* Have signs of infection (i.e., fever or current treatment with antibiotics)
* Have been exposed to an investigational drug/device within the preceding 30 days
* Be an employee of the site that is directly involved in the management, administration, or support of the study, or be an immediate family member of the same
* Be unwilling to or unable to comply with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
NEI score for Total Corneal Fluorescein Staining (TCFS) | 3 months
  To evaluate the efficacy of EBI-005 5 mg/mL topical ophthalmic solution given three times daily for 12 weeks as measured by the change in the NEI score for the Total Corneal Fluorescein Staining [sign] from baseline to Week 12 and a change in ocular pain as measured by the painful or sore eye question on the OSDI [symptom] of DED from baseline to Week 12 as compared to vehicle control.

SECONDARY OUTCOMES:
The key secondary endpoint is total OSDI score | 3 months
  Change from baseline to week 12 in Total OSDI score.

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Investigational Site, Chandler, Arizona
  - Investigational Site, Mesa, Arizona
  - Investigational Site, Little Rock, Arkansas
  - Investigational Site, Artesia, California
  - Investigational Site, Mission Hills, California
  - Investigational Site, Petaluma, California
  - Investigational Site, Rancho Cordova, California
  - Investiational Site, San Diego, California
  - Investigational Site, Torrence, California
  - Investigational Site, Littleton, Colorado
  - Investigational Site, Hamden, Connecticut
  - Investigational Site, Plantation, Florida
  - Investigational Site, Roswell, Georgia
  - Investigational Site, Bloomingdale, Illinois
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, New Albany, Indiana
  - Investigational Site, Lexington, Kentucky
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Bangor, Maine
  - Investigational Site, Boston, Massachusetts
  - Investigational Site, Winchester, Massachusetts
  - Investigational Site, Chesterfield, Missouri
  - Investigational Site, Des Peres, Missouri
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, St Louis, Missouri
  - Investigational Site, Washington, Missouri
  - Investigational Site, Las Vegas, Nevada
  - Investigational Site, New York, New York
  - Investigational Site, Rochester, New York
  - Investigational Site, Wantagh, New York
  - Investigational Site, High Point, North Carolina
  - Investigational Site, Cleveland, Ohio
  - Investigational Site, Cranberry Township, Pennsylvania
  - Investigational Site, Lancaster, Pennsylvania
  - Investigational Site, Pittsburgh, Pennsylvania
  - Investigational Site, Rapid City, South Dakota
  - Investigational Site, Memphis, Tennessee
  - Investigational Site, Houston, Texas
  - Investigational Site#2, Houston, Texas
  - Investigational Site, League City, Texas
  - Investigational Site, San Antonio, Texas
  - Investigational Site# 2, San Antonio, Texas
  - Investigational Site, Norfolk, Virginia